CLINICAL TRIAL: NCT00507182
Title: Fluorescence and Reflectance Spectroscopy for Diagnostic Assessment of Oral Mucosal Lesions
Brief Title: Spectroscopy for Diagnostic Assessment of Oral Mucosal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HNS99-100; NCI-2012-01601 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Oral Cancer
Keywords: Oral Mucosa Lesions; Oral Cancer; Neoplasia and Dysplasia in oral cavity mucosa; Fluorescence Spectroscopy; Reflectance Spectroscopy; Pre-cancerous lesions; Cancerous lesions; Mouth
MeSH Terms: conditions — Mouth Neoplasms; Neoplasms | interventions — Spectrometry, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorescence Spectroscopy (Experimental): 1-5 lesions + several normal-looking areas inside the mouth exposed to a beam of light; exposed tissues will emit very small amounts of fluorescence (light) then will be removed.
  Interventions: Procedure: Fluorescence Spectroscopy

INTERVENTIONS:
Procedure: Fluorescence Spectroscopy — 1-5 lesions + several normal-looking areas inside the mouth exposed to a beam of light; exposed tissues will emit very small amounts of fluorescence (light) then will be removed.

SUMMARY:
The goal of this clinical research study is to test a new way to look for cancer and pre-cancerous tissue changes inside the mouth.

DETAILED DESCRIPTION:
Abnormal-looking areas (lesions) inside the mouth may be a sign of cancer or changes that may lead to cancer. These lesions may need to be removed. Researchers are looking for a practical way to tell early on whether these lesions are cancer or may become cancer. This study will test a technique called fluorescence spectroscopy, which is under research in this study.

Each patient may have 1 to 5 lesions and several normal-looking areas inside the mouth exposed to a beam of light. The exposed tissues may emit very small amounts of light called fluorescence. This light is not seen by the eye but is detected by a computer. The small areas exposed to the light beam may then be removed.

The patients who need surgery may have the small tested areas removed when the lesions are surgically removed. A small sample from a normal-looking area may also be removed during surgery. Patients who do not need surgery may simply have small samples taken from the lesions and a normal-looking area in the clinic rather than in the operating room. The tissues will be looked at under a microscope to see whether they are cancerous. These results will be compared with the spectroscopy results.

If you are scheduled to participate in another MD Anderson study, Protocol 2008-0137 Entitled, "Phase Ib Study of Erlotinib Prior to Surgery in Patients with Head and Neck Cancer" (Study Chair: Dr. William William), some of your collected tissue samples may be shared with Dr. William for use on 2008-0137.

This is an investigational study. About 395 patients will be consented and screened for this study, with about 381 to take full part in this study. All will be treated at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Any person 18 years of age or older with a lesion of the oral mucosa. Persons with changes in existing lesions or those who develop new lesions can be re-evaluated, but it is not required.

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 1999-07-02 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Classification of Oral Lesions | 11 Years
  Distinguishing between normal and abnormal sites with four lesion classifications of normal, non-malignant inflammatory, dysplasia, and neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org